

Department of Psychiatry
University of California San Diego

9500 Gilman Drive La Jolla, CA 92093

## ACCESS TO TAILORED AUTISM INTEGRATED CARE PILOT STUDY

Document Date: 12/2/2020 (approval date)

NCT04293627

## **INFORMATION SHEET**

Adapting and Implementing an Integrated Care Model for Youth with Autism Spectrum Disorder and Psychiatric Comorbidity (Providers)

SPONSOR: National Institutes of Health INVESTIGATOR: Nicole Stadnick, PhD, MPH (858) 966-7703 x247101 EMAIL: ATTAIN@ucsd.edu

You are being invited to participate in a pilot study of the <u>Access To Tailored Autism IN</u>tegrated Care (ATTAIN) model. The purpose of this informational sheet is to provide you with information about this study.

- ➤ The purpose of this pilot study is to test the feasibility and acceptability of ATTAIN model, a refined way to improve identification of mental health problems and enhance referral to mental health care for children with autism spectrum disorder (ASD).
- > You are being asked to take part in this study because you are a pediatric provider caring for children with ASD.
- Participation in this study is entirely voluntary. You may choose not to be in this study. The data collected will not be shared with your employer, cannot be used for employee evaluation and will not affect your standing with your employer.
- You will be asked to participate in a 30-minute to one-hour training in the ATTAIN delivery process in advance of active implementation in your care setting. During this training, you will be asked to complete a brief 10-15-minute baseline survey about your background and attitudes towards using new innovations. You will receive a \$10 gift card for completing this survey.
- Over the course of 1 month, you will be asked to use or support use of the ATTAIN model with up to 5 eligible patients. Eligible patients are those who have a documented ASD diagnosis in their medical record, are between ages 4-16 years and speak English or Spanish. At the conclusion of 1 month, you will be asked to complete a brief 20-30-minute online survey regarding your experience using ATTAIN. You will receive a \$20 gift card for completing this survey.
- ➤ There are minimal risks if you participate in this study. Some of the questions may be considered sensitive, may be difficult to answer, or may cause uncomfortable feelings. You may refuse to answer any question.
- ➤ There is no guarantee that you will directly benefit from participating in this study. However, results from this research have the potential to benefit implementation of improved mental health screening and enhanced referral in pediatric primary care for children with ASD.
- The information collected will be shared only with the research team and will be kept strictly confidential.

If you have any questions about this study please contact:

Nicole Stadnick, PhD, MPH Principal Investigator University of California, San Diego (858) 966-7703 x247101; ATTAIN@ucsd.edu

If you have any questions about your rights as a research subject, please contact:

University of California, San Diego Human Research Protections Program (858) 246-4777

